CLINICAL TRIAL: NCT03101384
Title: Influence of Diagnostic Errors on the Prognosis of Acute Pulmonary Embolism
Acronym: IDEA-PE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: European Georges Pompidou Hospital (Other)
Responsible Party: Principal Investigator, Guy Meyer, Professeur des Universités, European Georges Pompidou Hospital
Other Study IDs: N° ID RCB : 2017-A00433-50
Record Dates: First submitted 2017-03-29; First posted 2017-04-05 (Actual); Last update posted 2017-06-02 (Actual); Status verified 2017-06

CONDITIONS: Pulmonary Embolism; Pulmonary Embolism and Thrombosis; Diagnostic Errors; Embolism; Pulmonary Vascular Disorder
MeSH Terms: conditions — Pulmonary Embolism; Thrombosis; Embolism | interventions — Diagnostic Errors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient with a diagnostic error: Defined by one of :
  1. Absence of prescribed test included in an accepted pulmonary diagnosis algorithm in the next 48h00 after the firts contact with a physician
  2. Absence of prescribed test included in an accepted pulmonary diagnosis algorithm by the first contacted physician but the diagnostic is done before 48h00 because the patient went at the emergency room on his own initiative.
  3. More than one doctor consulted before the diagnostic of pulmonary embolism (excluding the emergency physician if the patient was referred by the 1st contact doctor)
  Interventions: Other: Diagnostic error
- Patient without a diagnostic error: Any patient that did not meet the criteria to define the diagnostic error

INTERVENTIONS:
Other: Diagnostic error — There is no intervention in our study. Patient will be managed with usual care. We will divide patients in the 2 groups according to the presence of diagnostic error.
  Groups: Patient with a diagnostic error

SUMMARY:
Diagnostic errors have been reported frequently in patient with pulmonary embolism since symptoms are not specific. However, there is only scarce evidence that the delay associated with diagnostic errors may impact patient prognosis. The aim of this study is to determine the frequency of diagnostic errors and if they are associated with more severe pulmonary embolism in term of initial presentation and complications.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Episode of symptomatic acute pulmonary embolism objectively proven

Exclusion Criteria:

* Below 18 years of age
* Patient chronically receiving therapeutic anticoagulation
* Pulmonary embolism complicating a current hospitalisation for another medical reason
* Asymptomatic pulmonary embolism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with an episode of first acute symptomatic pulmonary embolism
Sampling Method: Non-Probability Sample
Enrollment: 302 (Estimated)
Dates: Start 2017-04-11 (Actual); Primary Completion 2018-10 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Severity of pulmonary embolism at the time of diagnosis | Day 1
  According to the 2014 Europe Society of Cardiology classification that combine clinical characteristics, signs of right ventricular dysfunction on imaging test and cardiac laboratory biomarkers

SECONDARY OUTCOMES:
Complication of pulmonary embolism | Day 30 and 180
  Composite of death, shock and recurrence
Frequency of diagnostic errors | Day 1
  Frequency of diagnostic errors
Characteristic of patient with diagnosis errors | Day 30
  Characteristic of patient with diagnosis errors

CONTACTS AND LOCATIONS:
Overall Officials: Guy Meyer, Pr, Principal Investigator — Hôpital Européen Georges Pompidou, AP-HP
Locations (1):
- Hôpital européen Georges Pompidou, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Undecided